CLINICAL TRIAL: NCT01370356
Title: A Phase 4, Multi-National, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of Varenicline Compared To Placebo For Smoking Cessation Through Reduction
Brief Title: A Study To Evaluate The Efficacy And Safety Of Varenicline Compared To Placebo For Smoking Cessation Through Reduction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: A3051075; REDUCE TO QUIT
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Smoking Cessation
Keywords: smoking reduction; smoking cessation
MeSH Terms: conditions — Smoking Cessation; Smoking Reduction | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline Tartrate (Active Comparator)
  Interventions: Drug: Varenicline Tartrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline Tartrate — Varenicline Tartrate oral tablets 2 (0.5mg) tablets twice a day for 24 weeks (first week titration)
  Arms: Varenicline Tartrate
Drug: Placebo — Matching placebo 2 oral tablets twice a day for 24 weeks (first week titration)
  Arms: Placebo

SUMMARY:
This study will determine whether varenicline is safe and helps people to quit smoking through reduction when they are not willing/able to make an abrupt quit attempt.

ELIGIBILITY:
Inclusion Criteria:

* Male and female cigarette smokers over the age of 18 years who are not willing/able to quit smoking within the next month but who are willing to attempt to reduce their smoking to work toward a quit attempt within the next 3 months.
* Subjects must have smoked an average of at least 10 cigarettes per day during the past year and during the month prior to the screening visit, with no continuous period of abstinence greater than 3 months in the past year and who have an exhaled carbon monoxide (CO) >10 ppm at screening.
* Subjects with mild to moderate depression or anxiety may be included if their condition is stable.

Exclusion Criteria:

* Subjects with a history of a suicide attempt or any suicidal behavior in the past two years.
* Subjects with severe depression or anxiety.
* Subjects with psychosis, panic disorder, bipolar disorder, post traumatic stress disorder (PTSD), or schizophrenia.
* Subjects with alcohol or substance abuse or dependence (except nicotine) unless in full remission for at least 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1510 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (65):
- United States (14):
  - Pharmacology Research Institute, Encino, California
  - Pharmacology Research Institute, Newport Beach, California
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CRI Worldwide, LLC, Marlton, New Jersey
  - Clinical Research Integrity(CRI) Worldwide, LLC, Willingboro, New Jersey
  - Central New York Clinical Research, Manlius, New York
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - Benchmark Research, Fort Worth, Texas
  - Healthfirst Medical Group, Fort Worth, Texas
- Australia (4):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Brisbane South Clinical Research Centre, Carina Heights, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Emeritus Research, Malvern, Victoria
- Canada (6):
  - Office of Dr. Ronald Collette, Burnaby, British Columbia
  - James K. Lai, MD., Inc., Vancouver, British Columbia
  - White Hills Medical Clinic, St. John's, Newfoundland and Labrador
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - Clinique des Maladies Lipidiques de Quebec (CMLQ), Québec, Quebec
- Czechia (7):
  - SurGal Clinic s.r.o., Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Krajska nemocnice Liberec a.s., Plicni oddeleni, Liberec
  - Mestska nemocnice Ostrava, Plicni oddeleni, Ostrava
  - Vseobecna fakultni nemocnice v Praze, III. interni klinika, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Ustredni vojenska nemocnice Praha, Prague
- Egypt (3):
  - Alexandria University, Alexandria
  - Ain Shams University Hospital, Cairo
  - El Fayoum university hospital, El Fayoum Qesm
- Germany (7):
  - Klinische Forschung Berlin, Berlin
  - Klinische Forschung Berlin-Buch GmbH, Berlin
  - Universitaetsklinikum Goettingen Zentrum Innere Medizin Abteilung Kardiologie und Pneumologie, Göttingen
  - Universitaetsklinikum Goettingen, Zentrum Innere Medizin, Abteilung Kardiologie und Pneumologie, Göttingen
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Medamed- Studienambulanz, Leipzig
  - FOCUS Clinical Drug Development GmbH, Neuss
- Japan (6):
  - Kubo Clinic, Yokohama, Kanagawa
  - Nagatsuta family clinic, Yokohama, Kanagawa
  - Sakakibara Clinic, Wakaumekai Medical Corporation, Yokohama, Kanagawa
  - Saino Clinic, Tokorozawa, Saitama
  - Tajima Clinic, Edogawa-ku, Tokyo
  - Hachiouji Junkanki clinic, Hachiōji, Tokyo
- Mexico (4):
  - Arke Estudios Clinicos S.A., México, D.f.
  - Centro Respiratorio de Mexico S.C., México, D.f.
  - Clinica de Enfermedades Cronicas y de Procedimientos Especiales S.C., Morelia, Michoacán
  - Centro de Estudios Clinicos y Especialidades Medicas SC, Monterrey, Nuevo León
- Taiwan (7):
  - Taichung Veterans General Hospital, Taichung, Taiwan
  - Chang Gung Medical Foundation-Linkou Branch, Kweishan Town, Taoyuan County
  - Kaohsiung Veterans General Hosptial, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Department of Family Medicine, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (7):
  - Enchord Limited, Fowey, Cornwall
  - The Alverton Practice, Penzance, Cornwall
  - Knowle House Surgery, Plymouth, Devon
  - Castlemilk Health Centre, Castlemilk, Glasgow
  - Prince Philip Hospital, Dafen, Llanelli
  - Hathaway Medical Centre, Chippenham, Wilts
  - The Jenner Practice, London

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Nakamura M, Abe M, Ohkura M, Treadow J, Yu CR, Park PW. Efficacy of Varenicline for Cigarette Reduction Before Quitting in Japanese Smokers: A Subpopulation Analysis of the Reduce to Quit Trial. Clin Ther. 2017 Apr;39(4):863-872. doi: 10.1016/j.clinthera.2017.03.007. Epub 2017 Mar 30. PMID 28365035
- [Derived] Ebbert JO, Hughes JR, West RJ, Rennard SI, Russ C, McRae TD, Treadow J, Yu CR, Dutro MP, Park PW. Effect of varenicline on smoking cessation through smoking reduction: a randomized clinical trial. JAMA. 2015 Feb 17;313(7):687-94. doi: 10.1001/jama.2015.280. PMID 25688780
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051075&StudyName=A%20Study%20To%20Evaluate%20The%20Efficacy%20And%20Safety%20Of%20Varenicline%20Compared%20To%20Placebo%20For%20Smoking%20Cessation%20Through%20Reduction

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1747 participants were screened, whereof 1510 were randomized into the study, and of whom 1493 took at least 1 dose of study drug. Overall, 61 centers in 10 countries received study drug: Australia (4), Canada (6), Czech Republic (6), Germany (6), Egypt (3), United Kingdom (7), Japan (6), Mexico (4), Taiwan (7), and USA (12).
Groups:
- Varenicline: Varenicline was titrated to the full dose during the first week (Day 1 - 3: 0.5 mg/day; Day 4 -7: 0.5 mg twice daily [BID]). From Week 2 to Week 24, the dose was 1 mg BID. Participants who had difficulties with tolerability were permitted to have the dose lowered temporarily or permanently to 0.5 mg BID. Data below are presented for the treated population.
- Placebo: Placebo was titrated and administered in the same manner as varenicline and reduction of dosing for difficulties with tolerability was also allowed. Data below are presented for the treated population.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 751 | 742
Completed | 559 | 515
Not Completed | 192 | 227
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 6 | 28
Not completed — Lost to Follow-up | 76 | 81
Not completed — Withdrawal by Subject | 54 | 59
Not completed — Reason not specified | 39 | 43
Not completed — Protocol Violation | 3 | 3
Not completed — Adverse event (AE) Related to Study Drug | 12 | 9
Not completed — AE Not Related to Study Drug | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Varenicline: Varenicline was titrated to the full dose during the first week (Day 1 - 3: 0.5 mg/day; Day 4 -7: 0.5 mg BID). From Week 2 to Week 24, the dose was 1 mg BID. Participants who had difficulties with tolerability were permitted to have the dose lowered temporarily or permanently to 0.5 mg BID. One participant was assigned to varenicline as a male but is in fact female. Data below are presented for the treated population.
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 751 | 742 | 1493
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (11.8) | 44.4 (12.0) | 44.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 330 | 321 | 651
  Male | 421 | 421 | 842

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Carbon Monoxide (CO) Confirmed 10-Week Continuous Abstinence (CA) From Smoking
Description: Percentage of participants who remained abstinent from Week 15 to Week 24, inclusive, reporting no smoking and no use of nicotine-containing products since the last study visit or contact on the Nicotine Use Inventory (NUI) and confirmed by expired CO < 10 ppm at any time point (CO measurements conducted at the clinic visits) during Weeks 15 through 24, inclusive. Missing CO was imputed as negative (CO ≤ 10 ppm).
Time Frame: Week 15 - 24
Population: The Full Analysis Set was referred to as the Intent-to-Treat (ITT) population and was defined as all randomized participants. The ITT population was the primary analysis set for the efficacy analyses in this study.
Measure: Number; unit: percentage of participants
Groups:
- Varenicline: Varenicline was titrated to the full dose during the first week (Day 1 - 3: 0.5 mg/day; Day 4 -7: 0.5 mg BID). From Week 2 to Week 24, the dose was 1 mg BID. Participants who had difficulties with tolerability were permitted to have the dose lowered temporarily or permanently to 0.5 mg BID.
- Placebo: Placebo was titrated and administered in the same manner as varenicline and reduction of dosing for difficulties with tolerability was also allowed.
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 760 | 750
percentage of participants | 32.1 | 6.9
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Assuming true CA rate of 6.9% for placebo and 17.2% for varenicline (odds ratio ≥ 2.8), a study randomizing 1404 participants (1:1 ratio) has ≥90% power to detect a difference between the two groups. Analysis was done using a logistic regression model; treatment effect as explanatory variable and investigative center as covariate. The interaction effect was tested using an expanded logistic regression model including treatment-by-center interaction; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical test was 2-sided and a 0.05 level of significance was used. A fixed-sequence procedure was used to adjust for multiplicity. Hierarchy of comparisons: 1) 10-week CA for Weeks 15 - 24, 2) CA for Weeks 21 - 24, 3) CA for Weeks 21 - 52; Odds Ratio (OR) = 8.74, 95% CI 2-sided [6.09 to 12.53]

2. Secondary Outcome: Percentage of Participants With CO Confirmed 4-Week CA From Smoking
Description: Percentage of participants who remained abstinent from Week 21 to Week 24, inclusive, reporting no smoking and no use of nicotine-containing products since the last study visit or contact on the NUI and confirmed by expired CO < 10 ppm at any time point (CO measurements conducted at the clinic visits) during Weeks 21 through 24, inclusive. Missing CO was imputed as negative (CO ≤ 10 ppm).
Time Frame: Week 21 - 24
Population: The Full Analysis Set was referred to as the ITT population and was defined as all randomized participants. The ITT population was the primary analysis set for the efficacy analyses in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 760 | 750
percentage of participants | 37.8 | 12.5
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Analysis was done using a logistic regression model including treatment effect as the explanatory variable and investigative center as covariate. In addition, the interaction effect was tested using an expanded logistic regression model including the treatment-by-center interaction. However, the inferences reported were based on the logistic regression model including only the main effects of treatment and center, regardless of the significance of the treatment by center interaction; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.66, 95% CI 2-sided [4.21 to 7.61]

3. Secondary Outcome: Percentage of Participants With CO Confirmed Long Term CA From Smoking
Description: Percentage of participants who remained abstinent from Week 21 to Week 52, inclusive, reporting no smoking and no use of nicotine-containing products since the last study visit or contact on the NUI and confirmed by expired CO < 10 ppm at any time point (CO measurements conducted at the clinic visits) during Weeks 21 through 52, inclusive. Missing CO was imputed as negative (CO ≤ 10 ppm).
Time Frame: Weeks 21 - 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 760 | 750
percentage of participants | 27.0 | 9.9
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.02, 95% CI 2-sided [2.94 to 5.50]

4. Secondary Outcome: Percentage of Participants With 7-Day Point Prevalence of Smoking Cessation
Description: The 7-day point prevalence of abstinence was defined as being abstinent from smoking and using tobacco products during the last 7 days at Week 12, 24, and 52. The participant's smoking status and other nicotine use was evaluated based on the "last 7 days" questions on the NUI and confirmed by CO expiration. Responders were defined as those, who answered "no" to both questions ("Has the subject smoked any cigarettes (even a puff) in the last 7 days?"; and "Has the subject used any nicotine products and/or other tobacco.... in the last 7 days?") and whose expired CO < 10 ppm. Missing CO was imputed as negative (CO ≤ 10 ppm).
Time Frame: Week 12, 24, and 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 760 | 750
percentage of participants
  Week 12 | 31.2 | 6.7
  Week 24 | 43.2 | 17.5
  Week 52 | 34.1 | 18.3
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Statistical analysis presented above is for Week 12. Analysis was done using logistic regression model with treatment effect as the explanatory variable and investigative center as covariate. The interaction effect was tested using an expanded logistic regression model with treatment-by-center interaction. The inferences reported were based on the logistic regression model including only the main effects of treatment and center, regardless of the significance of treatment by center interaction; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical test was 2-sided and a 0.05 level of significance was used; Odds Ratio (OR) = 8.69, 95% CI 2-sided [6.03 to 12.51]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Statistical analysis presented above is for Week 24. Analysis was done using logistic regression model with treatment effect as the explanatory variable and investigative center as covariate. The interaction effect was tested using an expanded logistic regression model with treatment-by-center interaction. The inferences reported were based on the logistic regression model including only the main effects of treatment and center, regardless of the significance of treatment by center interaction; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical test was 2-sided and a 0.05 level of significance was used; Odds Ratio (OR) = 4.58, 95% CI 2-sided [3.51 to 5.98]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Statistical analysis presented above is for Week 52. Analysis was done using logistic regression model with treatment effect as the explanatory variable and investigative center as covariate. The interaction effect was tested using an expanded logistic regression model with treatment-by-center interaction. The inferences reported were based on the logistic regression model including only the main effects of treatment and center, regardless of the significance of treatment by center interaction; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical test was 2-sided and a 0.05 level of significance was used; Odds Ratio (OR) = 2.66, 95% CI 2-sided [2.05 to 3.44]

5. Secondary Outcome: Percentage of Participants With 4-Week Point Prevalence of Smoking Cessation
Description: The 4-week point prevalence of abstinence was defined as being abstinent from smoking and using tobacco products during the last 4 weeks of the study. The participant's smoking status and other nicotine use was evaluated based on the "last 4 weeks" questions on the NUI and confirmed by CO expiration. Responders were defined as those, who answered "no" to both questions ("Has the subject smoked any cigarettes (even a puff) in the last 4 weeks?"; and "Has the subject used any nicotine products and/or other tobacco.... in the last 4 weeks?") and whose expired CO < 10 ppm. Missing CO was imputed as negative (CO ≤ 10 ppm).
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 760 | 750
percentage of participants | 32.8 | 17.3
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical test was 2-sided and a 0.05 level of significance was used; Odds Ratio (OR) = 2.67, 95% CI 2-sided [2.05 to 3.47]

ADVERSE EVENTS:
Time Frame: All AEs (serious and nonserious) were recorded from the date of first dose of study drug (Baseline) up to 30 days after the date of last dose of study drug.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 28/751 | 16/742
Other Adverse Events (participants affected / at risk) | 467/751 | 339/742
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=751) | Placebo (N=742)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Delirium tremens (Psychiatric disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0
Ovarian haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=751) | Placebo (N=742)
Constipation (Gastrointestinal disorders) | 38 | 13
Nausea (Gastrointestinal disorders) | 209 | 67
Fatigue (General disorders) | 46 | 34
Irritability (General disorders) | 39 | 30
Nasopharyngitis (Infections and infestations) | 98 | 89
Upper respiratory tract infection (Investigations) | 63 | 63
Headache (Nervous system disorders) | 62 | 54
Abnormal dreams (Psychiatric disorders) | 86 | 43
Anxiety (Psychiatric disorders) | 52 | 65
Insomnia (Psychiatric disorders) | 80 | 51

LIMITATIONS AND CAVEATS:
Two cases of fetal exposure during pregnancy occurred but are not included in the SAE section as they did not meet the criteria of serious in the safety database. One of them relates to a non-study participant who was the study participant's partner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.